CLINICAL TRIAL: NCT03105752
Title: Evaluation of the Readability of Information and Consent Forms on the Understanding of the Information Received by Participants in Biomedical Research
Brief Title: Evaluation of Readability of Consent Forms on the Understanding of the Information Received by Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIC-1421-14-02
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Outcome Assessments (Health Care); Comprehension; Language
Keywords: Outcome Assessments (Health Care); Volunteers; Informed consent; Comprehension; Language tests
MeSH Terms: conditions — Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Research participants (Experimental): Each participant of a clinical trial completed the "Qualité de Compréhension des Formulaires d'information et de consentement" questionnaire (QCFic) about its understanding of the information received. This questionnaire was retrieved immediately on the day of consent, with no possibility of referring to the content of information letter.
  Interventions: Other: Questionnaire of understanding

INTERVENTIONS:
Other: Questionnaire of understanding — The study involved 12 clinical trials conducted in the Clinical Research Center Paris Est. Twenty participants per trial were offered to answer the "Qualité de Compréhension des Formulaires d'information et de consentement" questionnaire (QCFic) at the inclusion visit after receiving the information by the investigator and signed or refused to sign the form of consent.
  Participants filled out the questionnaire in an isolated location, with no possibility of re-reading the information contained in the consent form. The questionnaire was immediately retrieved.

SUMMARY:
Prior to the completion of biomedical research, any person undergoing it must receive a readable and intelligible information about this research, in order to give free and informed consent. The willingness to inform patients of all risks and constraints related to research may be in contradiction with the need to write informative and concise documents that are understandable to research participants. As a result, consent forms are long, contain a lot of information and are complicated to understand.

The objective of this study is to evaluate the impact of the readability of the information and consent forms on the understanding of the information received by participants in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Every volunteers included in a study in a french clinical research center
* Ability to read and write in French

Exclusion Criteria:

* Refusal of participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the overall comprehension score and the readability index of Flesch | Immediate evaluation

SECONDARY OUTCOMES:
Correlation between the overall comprehension score and the level of education | Immediate evaluation
Correlation between the overall comprehension score and the status of volunteer | Immediate evaluation
Correlation between the overall comprehension score and the type of study | Immediate evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Funck-Brenta, MD, PhD, Study Director — Centre d'investigation clinique Paris Est

IPD SHARING:
Plan to Share IPD: No